CLINICAL TRIAL: NCT06434961
Title: A Multicenter, Randomised, Double-blind, Double-dummy Study to Assess the Efficacy and Safety of SHR6508 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Brief Title: The Trial of SHR6508 in Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR6508-301
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: SHR6508 plus oral placebo tablets
- Active Control group (Active Comparator)
  Interventions: Drug: Cinacalcet plus intravenous placebo

INTERVENTIONS:
Drug: SHR6508 plus oral placebo tablets — SHR6508 plus oral placebo tablets
  Arms: Treatment group
Drug: Cinacalcet plus intravenous placebo — Cinacalcet plus intravenous placebo
  Arms: Active Control group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR6508 among Chinese patients with secondary hyperparathyroidism of chronic kidney disease treated by maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Diagnosed with end stage renal disease receiving maintenance hemodialysis
3. Male or female
4. Meet the Body Mass Index standard
5. Stably use of concomitant medication of other therapies of SHPT
6. Meet the standard of iPTH level, cCa

Exclusion Criteria:

1. Subjects with a history of malignant tumor
2. Subjects with neuropsychiatric diseases
3. Subjects with a history of cardiovascular diseases
4. Subjects with gastrointestinal diseases
5. Subjects with a history of surgery
6. Subjects with a history of blood loss
7. Abnormal blood pressure, serum magnesium, serum transaminase, serum albumin
8. Subjects with a treatment history of similar drugs
9. Allergic to a drug ingredient or component
10. Pregnant or nursing women
11. No birth control during the specified period of time
12. Subject with a history of alcohol abuse and drug abuse
13. Participated in clinical trials of other drugs
14. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants to End of Study whose iPTH decreased by>30% from baseline | efficacy assessment period, defined as Week 20-27
  iPTH was tested at a central laboratory.

SECONDARY OUTCOMES:
Proportion of Participants to End of Study whose iPTH decreased by>50% from baseline | efficacy assessment period, defined as Week 20-27
  iPTH was tested at a central laboratory.
Incidence of nausea and vomiting events | Day1 to End of Treatment, End of Treatment is about Week 27
  Terms were coded with Medical Dictionary for Regulatory Activities (MedDRA)
Proportion of Participants to End of Treatment whose iPTH decreased to 300 pg/mL from baseline | efficacy assessment period, defined as Week 20-27
  iPTH was tested at a central laboratory.
Change From Baseline in serum cCa and P | efficacy assessment period, defined as Week 20-27
  cCa and P were tested at a central laboratory.
Participants With Treatment-Emergent Adverse Events (TEAEs) | Day1 to End of Study, End of Study is about Week 31
  Terms were coded with Medical Dictionary for Regulatory Activities (MedDRA)
Participants with Anti-SHR6508 Antibody at baseline and postbaseline | Day1 to End of Study, End of Study is about Week 31
  Anti-SHR6508 Antibody was measured in patient serum samples using a validated enzyme-linked immunosorbent assay (ELISA) method.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided